CLINICAL TRIAL: NCT05227326
Title: First in Human Phase 1 Study of AOH1996 in Patients With Refractory Solid Tumors
Brief Title: AOH1996 for the Treatment of Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21310; NCI-2021-14102 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21310 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-02-07 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Refractory Malignant Solid Neoplasm; Osteosarcoma; Leiomyosarcomas; Synovial Sarcomas; Ovarian Cancer; Non-Small Cell Lung Cancer; Pancreatic Cancer
MeSH Terms: conditions — Osteosarcoma; Leiomyosarcoma; Sarcoma, Synovial; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (PCNA inhibitor AOH1996) (Experimental): Patients receive PCNA inhibitor AOH1996 PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PCNA Inhibitor AOH1996

INTERVENTIONS:
Drug: PCNA Inhibitor AOH1996 — Given PO
  Other Names: AOH 1996; AOH-1996; AOH1996; Proliferating Cell Nuclear Antigen Inhibitor AOH1996

SUMMARY:
This phase I trial studies the side effects and best dose of AOH1996 in treating patients with solid tumors that do not respond to treatment (refractory). AOH1996 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of AOH1996.

II. To establish the recommended phase 2 dose of AOH1996.

III. To establish the recommended phase 2 dose of AOH1996 when given in conjunction with a TKI for NSCLC.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics of AOH1996. II. To evaluate for preliminary efficacy of AOH1996. III. To evaluate response rate and disease control rate in solid tumors.

EXPLORATORY OBJECTIVE:

I. To determine pharmacodynamics parameters (alteration of gammaH2AX, downregulation of Myc) of AOH1996.

OUTLINE: This is a dose-escalation study.

Patients receive AOH1996 orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent and Willingness to Participate

* 1. Documented informed consent by the participant
* 2. Willingness to permit study team to obtain and use archival tissue, if already existing

Age Criteria, Performance Status and Life Expectancy

* 3. Age: ≥ 18 years
* 4. ECOG performance status ≤ 2
* 5. Life expectancy of > 3 months

Nature of Illness and Treatment History __6. Patients with solid tumors failing standard therapies or patients refusing standard treatments (exception: Part B NSCLC combination (EGFR TKI + AOH1996) cohort: patients with stable disease or better on EGFR TKI for at least 2 months)

Contraception

__7. Agreement by females and males of childbearing potential* to use an adequate method of birth control (hormonal contraception is inadequate) or abstain from heterosexual activity for the course of the study through 30 days after the last dose of study medication. See Appendix B for guidelines.

- Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Laboratory Criteria (to be performed within 14 days prior to Day 1)

* 8. ANC ≥ 1,500/mm3
* 9. Platelets ≥ 100,000/mm3 :
* 10. Total serum bilirubin ≤ 1.5 x ULN
* 11. AST =< 1.5 x ULN or =< 3 x ULN with liver metastases
* 12. ALT =< 1.5 x ULN or =< 3 x ULN with liver metastases
* 13. Creatinine clearance of ≥ 60 mL/min per 24 hour urine or the Cockcroft-Gault
* 14. Women of childbearing potential (WOCBP): negative urine or serum pregnancy test If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

Exclusion Criteria

Concomitant Medications/Therapies __1. Dietary/herbal supplements

* 2. Other investigational products or chemotherapy. Exception: EGFR TKI in the NSCLC expansion cohort is allowed.
* 3. Warfarin
* 4. Current or planned use of agents contraindicated for use with strong CYP3A4 inducers
* 5. Strong inhibitors or inducers of CYP2C9
* 6. Strong inhibitors or inducers of CYP3A

Other Illnesses and Conditions

* 7. Issues with tolerating oral medication (e.g., inability to swallow pills, malabsorption issues, ongoing nausea or vomiting).
* 8. Women who are or are planning to become pregnant or breastfeed
* 9. Known allergy to any of the components within the study agents and/or their excipients.
* 10. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years.
* 11. Intercurrent or historic medical condition that increases subject risk in the opinion of the Investigator. Eligibility may be revisited for intercurrent medical conditions once resolution/recovery is deemed adequate by the investigator (e.g. recovery from major surgery, completion of treatment for severe infection).

Noncompliance

__12. Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

**Eligibility should be confirmed per institutional policies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2029-09-13 (Estimated); Study Completion 2029-09-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last study drug is given
  Toxicity and adverse events will be recorded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All toxicities/AEs will be recorded from the initiation of protocol therapy through the follow-up period.
Dose limiting toxicities | Up to 28 days (cycle 1)
  Toxicities will be graded according to NCI CTCAE version 4.0.

SECONDARY OUTCOMES:
Response rate | Up to 2 years
  Will be assessed using Response Evaluation Criteria in Solid Tumors version 1. Response rate will be estimated in the overall population and 95% exact confidence intervals will be estimated.
Progression-free survival | Assessed up to 2 years
  Time to disease progression/ relapse or death as a result of any cause.
Overall survival | Assessed up to 2 years
  Time to death as a result of any cause.
Time to treatment failure | Assessed up to 2 years
  Time to treatment termination for any reason (progression, toxicity, death, patient preference).

OTHER OUTCOMES:
Levels of plasma gammaH2AX | Up to 2 years
  Will use descriptive statistics and graphical displays to summarize levels of plasma gammaH2AX, evaluate changes between pre- and post-treatment measurements. A paired t-test will be used to determine if there is a statistically significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - Honor Health Research and Innovation Institute, Scottsdale, Arizona
  - City of Hope Medical Center, Duarte, California